CLINICAL TRIAL: NCT05625854
Title: The Effect of Using a Fan With Aromatherapy in Breathlessness Patient in Terminally Illness: a Randomized Control Trial
Brief Title: Using a Fan With Aromatherapy in Breathlessness Patients in Terminal Illness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tsai-Wei Huang (Other)
Responsible Party: Sponsor-Investigator, Tsai-Wei Huang, Associate professor, Taipei Medical University
Organization: Taipei Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: fan for dyspnea
Record Dates: First submitted 2021-09-14; First posted 2022-11-23 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Breathlessness; Aromatherapy; Fans; Terminal Illness
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Blow a fan to the face combine aromatherapy (Experimental)
  Interventions: Behavioral: Blow a fan to the face combine aromatherapy
- Blow a fan to the face (Experimental)
  Interventions: Behavioral: Blow a fan to the face
- Blow a fan to the feet (Placebo Comparator)
  Interventions: Behavioral: Blow a fan to the feet

INTERVENTIONS:
Behavioral: Blow a fan to the face combine aromatherapy — Blow a fan with aromatherapy to the face
  Arms: Blow a fan to the face combine aromatherapy
Behavioral: Blow a fan to the face — Blow a fan to the face
  Arms: Blow a fan to the face
Behavioral: Blow a fan to the feet — Blow a fan to the feet
  Arms: Blow a fan to the feet

SUMMARY:
Difficulty breathing is a very devastating symptom, often seen in terminal patients. Accompanied by physical, psychological, emotional, and social limitations, Not to mention the ambiguity in the occurrence of dyspnea symptoms and the difficulty in obtaining satisfactory quality of symptom care. The purpose of this study is to confirm the use of non-drug interventions in clinical situations, such as fans and aromatherapy to alleviate the complications of end-stage patients. The effectiveness of the symptoms of dyspnea.

DETAILED DESCRIPTION:
Difficulty breathing is a very devastating symptom, often seen in terminal patients. Accompanied by physical, psychological, emotional, and social limitations, Not to mention the ambiguity in the occurrence of dyspnea symptoms and the difficulty in obtaining satisfactory quality of symptom care. The purpose of this study is to confirm the use of non-drug interventions in clinical situations, such as fans and aromatherapy to alleviate the complications of end-stage patients. The effectiveness of the symptoms of dyspnea.

Inclusion criteria

1. Over 20 years old.
2. It is determined by the physician to meet the final diagnosis conditions.
3. Symptoms of dyspnea.
4. The daily physical status of patients is assessed using the East Coast Cancer Clinical Research Cooperative Organization Assessment Scale (Eastern Cooperative Oncology Group, ECOG) ≧ 2 points.
5. Able to communicate in Mandarin or Taiwanese or written conversation.
6. Unconscious disorder.
7. After explaining and explaining, agree to participate in this research and sign the consent form.

Exclusion criteria

1. Receive treatment for facial trigeminal nerve damage.
2. Abnormal sense of smell.

ELIGIBILITY:
Inclusion Criteria:

1. Over 20 years old.
2. It is determined by the physician to meet the final diagnosis conditions.
3. Symptoms of dyspnea.
4. The status of patients is assessed using the East Coast Cancer Clinical Research Cooperative Organization Assessment Scale (ECOG) ≧ 2 points.
5. Able to communicate in Mandarin or Taiwanese or written conversation.
6. Conscience clear.
7. After explaining and explaining, agree to participate in this research and sign the consent form.

Exclusion Criteria:

1. Receive treatment for facial trigeminal nerve damage.
2. Abnormal sense of smell.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2022-11-25 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Chinese version of the Respiratory Distress Observation Scale，C-RDOS | The score change up to three days.
  RDOS is an eight-item ordinal scale designed to measure the presence and intensity of respiratory distress in adults. High score means high respiratory distress.

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | The score change up to three days.
  The PHQ-9 is the depression module, which scores each of the nine DSM-IV criteria as "0" (not at all) to "3" (nearly every day). It has been validated for use in primary care.[2]
  It is not a screening tool for depression but it is used to monitor the severity of depression and response to treatment. high score mean higher emotion distress.
Chinese version of the Edmonton Symptom Assessment System，C-ESAS | The score change up to three days.
  The ESAS includes 11 symptoms: pain, tiredness, nausea, depression, anxiety, drowsiness, appetite, sleep, well-being, shortness of breath, and other. It uses a 0-10 numerical scale: 0 shows the absence of a symptom, and 10 shows the worst experience of the symptom.
Smart bracelet_Heart rate variability (HRV) | Continue wear bracelet five days to record HRV data.
  HRV is the physiological phenomenon of the variation in the time interval between consecutive heartbeats in milliseconds. A normal, healthy heart does not tick evenly like a metronome, but instead, when looking at the milliseconds between heartbeats, there is constant variation.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University, Taipei, Taiwan